CLINICAL TRIAL: NCT06042894
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of SI-B003 Monotherapy or BL-B01D1+SI-B003 Combination Therapy (BL-B01D1+SI-B003) in Patients With Unresectable Locally Advanced or Recurrent Metastatic HER2 Negative Breast Cancer
Brief Title: A Study of SI-B003 or BL-B01D1+SI-B003 in Patients With Unresectable Locally Advanced or Recurrent Metastatic HER2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-SI-B003-201-04
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: HER-2 negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 + SI-B003 (Experimental): Participants receive SI-B003 or BL-B01D1 + SI-B003 therapy in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-B01D1; Drug: SI-B003

INTERVENTIONS:
Drug: BL-B01D1 — BL-B01D1 was administered by intravenous infusion on D1 and D8 in a 3-week cycle.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: SI-B003 — SI-B003 was administered by intravenous infusion on D1 in a 3-week cycle.

SUMMARY:
This phase II study is a clinical study to explore the efficacy and safety of SI-B003 monotherapy and BL-B01D1+SI-B003 combination therapy in patients with unresectable locally advanced or recurrent metastatic HER-2 negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol.
2. Age: ≥18 years old and ≤75 years old.
3. Expected survival time ≥3 months.
4. ECOG 0 or 1.
5. Pathologically and/or cytologically confirmed patients who have failed standard treatment, or have no access to standard treatment Patients with unresectable, locally advanced or recurrent, metastatic HER2-negative breast cancer after posterior line.
6. Agree to provide archived tumor tissue specimens (unstained sections (anti-slip)) from primary or metastatic sites within 2 years. 10 to 12 surgical specimens (4-5 μm thick) or fresh tissue samples if the subject is unable to provide them for 2 years tumor tissue samples from within, can be communicated with the sponsor if other inclusion criteria are met, enrollment was permitted after investigator assessment.
7. Must have at least one measurable lesion according to RECIST v1.1 definition; So let's say that we've done this before radiotherapy-treated lesions were included only if there was definite disease progression in the lesion after radiotherapy measurable lesions were entered.
8. Blood transfusions, the use of any cell growth factors, and/or blood transfusions were not allowed within 14 days before screening in the presence of a platelet drug, the organ function level must meet the following criteria:

   1. Blood routine: hemoglobin (HGB) ≥ 90g/L; Absolute neutrophil count (NEUT) ≥ 1.5× 10 9 /L; Platelet count (PLT) ≥ 90× 10 9 /L;
   2. Renal function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (According to Cockcroft and Gault formula);
   3. Liver function: total bilirubin (TBIL≤1.5 ULN), alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) was ≤2.5 ULN in all patients, and AST and ALT were ≤ in patients with liver metastasis 5.0 ULN;
   4. Coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5ULN;
   5. no severe cardiac dysfunction with left ventricular ejection fraction ≥50%;
   6. proteinuria ≤2+ or ≤1000mg/24h.
9. Toxicity from previous antineoplastic therapy has returned to grade 1 or less as defined by NCI-CTCAE v5.0 (investigator review) concerns about asymptomatic laboratory abnormalities such as elevated ALP, hyperuricemia, hyperglycemia, etc., and investigators toxicity without safety risk was judged, such as alopecia, grade 2 peripheral neurotoxicity, or decreased hemoglobin but ≥90g/L except).
10. A pregnancy test should be performed within 7 days of starting treatment for premenopausal women who are likely to have children clear or urine pregnancy tests must be negative and must be non-lactating; All enrolled patients should be in the entire treatment week adequate barrier contraceptive measures were taken at the end of treatment and 6 months after the end of treatment.

Exclusion Criteria:

1. ADC drugs that have received topoisomerase I inhibitors (camptothecins) as small molecule toxins.
2. Administration of chemotherapy or chemotherapy within 4 weeks or 5 half-lives, whichever is shorter, before the first dose physical therapy, immunotherapy, definitive radiotherapy, major surgery (investigator's definition), targeted therapy (including minor) molecular tyrosine kinase inhibitors) and other anti-tumor therapy; Oral fluorouracil drugs such as S-1, carboplatin ecitabine or palliative radiotherapy within 2 weeks before the first dose.
3. Use of immunomodulatory drugs within 14 days before the first use of the study drug: including but not limited to thymosin, interleukin-2, interferon, etc.
4. Systemic corticosteroids (> 10mg/ day prednisone, or other corticosteroids in equivalent amounts); Inhaled or topical administration of hormones, or received physiology for adrenal insufficiency alternative doses of hormone therapy were excluded.
5. Patients with grade ≥3 irAE or grade ≥2 immune-related myocarditis who had received immunotherapy were excluded.
6. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

   1. severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias or grade III atria requiring clinical intervention Ventricular block;
   2. prolonged QT interval at rest (QTc > 450 msec in men or QTc > 470 msec in women);
   3. myocardial infarction, unstable angina, cardiac angioplasty, or within 6 months before the first dose Stent implantation, coronary artery/peripheral artery bypass grafting, New York Heart Association Defined class III or IV congestive heart failure, cerebrovascular accident, or transient ischemic attack.
7. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, silver requiring systemic treatment dandruptitis, rheumatoid arthritis, inflammatory bowel disease and hashimoto's thyroiditis, except type I diabetes, hypothyroidism that can be controlled only by replacement therapy, skin diseases that do not require systemic treatment (e.g., vitiligo, silver) Dandruff).
8. Other malignancies that progressed or required treatment within 3 years before the first dose, such as the following external: radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or radical carcinoma in situ.
9. History or current history of (noninfectious) interstitial lung disease (ILD)/pulmonary inflammation requiring steroid therapy patients with ILD/ pulmonary inflammation, or suspected ILD/ pulmonary inflammation that cannot be excluded by imaging at the time of screening.
10. Prior to starting the study treatment, there are:

    1. Poorly controlled diabetes (fasting blood glucose ≥ 13.3 mmol/L)
    2. Poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
    3. History of hypertensive crisis or hypertensive encephalopathy.
11. Unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening thrombotic events such as plug; Infusion-related thrombosis was excluded.
12. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases). Patients who had received treatment for brain metastases (radiotherapy or surgery; Patients with stable brain metastases who had stopped radiotherapy or surgery 28 days before the first dose were eligible. Patients with cancerous meningitis (meningeal metastasis) were excluded even if they were treated and judged to be stable. Stability is defined as meeting the following four criteria:

    1. seizure-free status for > 12 weeks with or without antiepileptic medication;
    2. no need for corticosteroids;
    3. stable on two consecutive MRI scans (at least 4 weeks apart);
    4. stable and asymptomatic for more than one month after treatment.
13. Patients with pleural effusion, pericardial effusion or ascites with clinical symptoms or requiring repeated drainage.
14. Allergic history to recombinant humanized antibody or human-mouse chimeric antibody or any excipients of BL-B01D1 sensitive patients.
15. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
16. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > lower detection limit).
17. Positive hepatitis B surface antigen (HBsAg) and HBV DNA> 500IU/ml or 2000 copies /ml patients with HBV infection should receive antiviral treatment according to local treatment guidelines and be willing to participate in the study all patients received antiviral therapy during the whole period.
18. Active infection requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
19. Had participated in another clinical trial within 4 weeks before the first dose (calculated from the time of last dose).
20. Persons with a history of psychotropic drug abuse and inability to quit or mental disorders.
21. Any other circumstances that the investigator deemed inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study .

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, PHD, Principal Investigator — Fudan University; Jian Zhang, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China